CLINICAL TRIAL: NCT04899739
Title: Prospective Study of Preoperative Diagnostic Endoscopy for the Diagnosis of Occult Metastatic Lesions of Operable Pancreatic Cancer
Brief Title: Intraoperative Endoscopic Ultrasound for Pancreatic Cancer
Acronym: EchoSurg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-007
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
Keywords: EUS; Endoscopic Ultrasound; Biopsy; Pancreatic surgery; Pancreatic Cancer; Artificial intelligence
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peripancreatic and distant lymph node assessment (Experimental): All patients programmed for an endoscopic ultrasound in the context of a pancreatic cancer
  Interventions: Diagnostic Test: Echoendoscopy

INTERVENTIONS:
Diagnostic Test: Echoendoscopy — Peripancreatic lymph nodes and at a distance from the pancreas assessment by endoscopic ultrasound, elastography an doppler to record their anatomical location and characteristics. All lymph nodes suspected of metastatic disease will be marked with sterile black ink.

SUMMARY:
Nowadays pancreatic cancer is one of the deadliest oncological pathologies. The only effective curative tool is the surgery. Before the intervention, an endoscopic ultrasound is performed on the patient to carry out the biopsy of the main tumor. In this study, the echoendoscopie will be extended to lymph node staging away from the surgical field in order to implement a simple classification of lymph nodes, based on non-invasive ultrasound criteria. This would facilitate the location and qualification of peripancreatic lymph nodes and distant from the tumor, and therefore the staging of the tumor.

DETAILED DESCRIPTION:
Nowadays pancreatic cancer is one of the deadliest oncological pathologies today. Even after curative surgery, considered the only effective curative tool, 5-years survival does not exceed 5%. Before surgery, an endoscopic ultrasound is performed on the patient to carry out the biopsy of the main tumor. However, the evaluation being devoted to the pancreas, this study wishes to extend echoendoscopie to lymph node staging away from the surgical field. The proposed study is based on the hypothesis that the implementation of a simple classification of lymph nodes, based on non-invasive ultrasound criteria, would facilitate the location and qualification of peripancreatic lymph nodes and distant from the tumor, and therefore the staging of the tumor.

At the same time, the video data obtained will be collected in a computer database in order to create an artificial intelligence lesion detection and qualification tool.

This study plans to recruit 45 adult patients, male or female, with a solid or cystic pancreatic tumor and for whom a surgical resection (first line and after neoadjuvant treatment) is planned. The main objective is to estimate the sensitivity and specificity of a simple classification "benign / malignant" of the nodes, established by the endoscopist using endoscopic ultrasound criteria's, compared to the gold standard (anatomopathology).

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years old
2. Patient with a solid or degenerated cystic tumor of the pancreas requiring curative surgery
3. Patient with a complete clinical examination performed
4. Patient with no contraindication to anesthesia, upper digestive endoscopy and pancreatic surgery
5. Patient able to receive and understand information relating to the study and give informed written consent
6. Patient affiliated to the French social security system

Exclusion Criteria:

1. Patient presenting with bleeding disease with disorder hemostasis and coagulation (PT <60%, TCA> 40 s and platelets <60,000 / mm3)
2. Patient on anticoagulant or antiaggregant treatment that cannot be temporarily interrupted
3. Patient carrying a right-left shunt, a severe pulmonary arterial hypertension (high blood pressure pulmonary> 90 mm Hg), uncontrolled systemic hypertension or suffering from respiratory distress syndrome.
4. Pregnant or breastfeeding patient
5. Patient in exclusion period (determined by a previous study or in progress)
6. Patient under legal protection
7. Patient under guardianship or trusteeship

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of lymph nodes correctly categorised by ultrasound endoscopy. (Sensitivity) | 1 month
  Number of lymph nodes correctly categorised by ultrasound endoscopy compared to the gold standard (anatomopathology).
Rate of lymph nodes wrongly categorised by ultrasound endoscopy. (Specificity) | 1 month
  Number of lymph nodes wrongly categorised by ultrasound endoscopy compared to the gold standard (anatomopathology).

SECONDARY OUTCOMES:
Rate of metastases actually diagnosed | 1 month
  Comparison between the number of suspected lymph nodes identified during preoperative endoscopic ultrasound and results of the histological analysis of these resected lymph nodes.
Location of hidden lymph node metastases | 1 day
  Description of the location of hidden lymph node metastases identified by endoscopic ultrasound
Number of distant nodes detected during the endoscopic ultrasound | 1 day
  Number of distant nodes detected during the preoperative endoscopic ultrasound
Number of distant malignant lymph nodes | 1 month
  Number of distant lymph nodes detected during the preoperative endoscopic ultrasound and whose malignancy has been confirmed by the gold standard
Rate of patients for whom contraindications for surgery has been detected during the endoscopic ultrasound | 1 day
  Number of patients for whom a contraindication to surgery has been detected during the endoscopic ultrasound, on the total number of patients included.
Rate of patients for whom elastography was required to identify lymph node metastases hidden away from the surgical site | 1 day
  Number of patients for whom elastography was required to identify distant hidden lymph node metastases
Measurement of the operating time required to perform preoperative elastography | 1 day
  Measurement of the operating time (in minutes) required to perform preoperative elastography.
Measurement of the additional costs generated by materials required for preoperative elastography | 1 day
  Measurement of the additional costs (in euros) generated by materials required for preoperative elastography in resectable pancreas cancer patients
Impact of sterile black ink marking of distant nodes during the preoperative EA | 1 day
  Analysis of the impact of sterile black ink marking of distant lymph nodes during preoperative ultrasound endoscopy on the surgical procedure by the mean of a questionnaire completed by the surgeon. This questionnaire will be assessed by a score of Likert varying between 1 (not satisfied) and 5 (very satisfied).
Development of an algorithm capable of detecting lymph nodes metastases by the mean of artificial intelligence | 1 day
  Deep learning-based analysis of video data from the ultrasound endoscopy
Development of an algorithm capable of characterizing lymph nodes metastases by the mean of artificial intelligence | 1 day
  Deep learning-based analysis of video data from the ultrasound endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Pessaux, MD, Principal Investigator — Unité de Chirurgie Hépato-biliaire et Pancréatique, NHC Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Kleeff J, Reiser C, Hinz U, Bachmann J, Debus J, Jaeger D, Friess H, Buchler MW. Surgery for recurrent pancreatic ductal adenocarcinoma. Ann Surg. 2007 Apr;245(4):566-72. doi: 10.1097/01.sla.0000245845.06772.7d. PMID 17414605
- [Background] Poruk KE, Firpo MA, Adler DG, Mulvihill SJ. Screening for pancreatic cancer: why, how, and who? Ann Surg. 2013 Jan;257(1):17-26. doi: 10.1097/SLA.0b013e31825ffbfb. PMID 22895395
- [Background] Butturini G, Stocken DD, Wente MN, Jeekel H, Klinkenbijl JH, Bakkevold KE, Takada T, Amano H, Dervenis C, Bassi C, Buchler MW, Neoptolemos JP; Pancreatic Cancer Meta-Analysis Group. Influence of resection margins and treatment on survival in patients with pancreatic cancer: meta-analysis of randomized controlled trials. Arch Surg. 2008 Jan;143(1):75-83; discussion 83. doi: 10.1001/archsurg.2007.17. PMID 18209156
- [Background] Galasso D, Carnuccio A, Larghi A. Pancreatic cancer: diagnosis and endoscopic staging. Eur Rev Med Pharmacol Sci. 2010 Apr;14(4):375-85. PMID 20496552
- [Background] Al-Haddad M, Wallace MB, Woodward TA, Gross SA, Hodgens CM, Toton RD, Raimondo M. The safety of fine-needle aspiration guided by endoscopic ultrasound: a prospective study. Endoscopy. 2008 Mar;40(3):204-8. doi: 10.1055/s-2007-995336. Epub 2007 Dec 4. PMID 18058615
- [Background] Bhutani MS, Hawes RH, Hoffman BJ. A comparison of the accuracy of echo features during endoscopic ultrasound (EUS) and EUS-guided fine-needle aspiration for diagnosis of malignant lymph node invasion. Gastrointest Endosc. 1997 Jun;45(6):474-9. doi: 10.1016/s0016-5107(97)70176-7. PMID 9199903
- [Background] Kanamori A, Hirooka Y, Itoh A, Hashimoto S, Kawashima H, Hara K, Uchida H, Goto J, Ohmiya N, Niwa Y, Goto H. Usefulness of contrast-enhanced endoscopic ultrasonography in the differentiation between malignant and benign lymphadenopathy. Am J Gastroenterol. 2006 Jan;101(1):45-51. doi: 10.1111/j.1572-0241.2006.00394.x. PMID 16405532
- [Background] Giovannini M, Thomas B, Erwan B, Christian P, Fabrice C, Benjamin E, Genevieve M, Paolo A, Pierre D, Robert Y, Walter S, Hanz S, Carl S, Christoph D, Pierre E, Jean-Luc VL, Jacques D, Peter V, Andrian S. Endoscopic ultrasound elastography for evaluation of lymph nodes and pancreatic masses: a multicenter study. World J Gastroenterol. 2009 Apr 7;15(13):1587-93. doi: 10.3748/wjg.15.1587. PMID 19340900
- [Background] Nawaz H, Fan CY, Kloke J, Khalid A, McGrath K, Landsittel D, Papachristou GI. Performance characteristics of endoscopic ultrasound in the staging of pancreatic cancer: a meta-analysis. JOP. 2013 Sep 10;14(5):484-97. doi: 10.6092/1590-8577/1512. PMID 24018593